CLINICAL TRIAL: NCT07256197
Title: Effect and Safety of PCSK9 Inhibitors on the Progression of Mild/Middle Calcific Aortic Stenosis: A Randomized Controlled Clinical Trial
Brief Title: PCSK9 Inhibitors in the Treatment of Calcific Aortic Stenosis
Acronym: PICASO
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Anzhen Hospital (Other)
Collaborators: Beijing Jishuitan Hospital (Other); Chinese Academy of Medical Sciences, Fuwai Hospital (Other); Beijing Hospital (Other Government); Nanchong Central Hospital (Other Government); Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Zhi Jian Wang, Professor, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PICASO
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Aortic Stenosis, Calcific
Keywords: PCSK9 Inhibitors; Calcific Aortic Stenosis
MeSH Terms: conditions — Aortic Valve, Calcification of | interventions — Therapeutics; PCSK9 Inhibitors

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment with PCSK9 inhibitors (Experimental): Patients in experimental group are treated with PCSK9 inhibitors (150mg Tafolecimab subcutaneously every two weeks) and guideline-directed management in cardiovascular primary or secondary prevention.
  Interventions: Drug: Treatment with PCSK9 inhibitors
- Treatment without PCSK9 inhibitors (Other): Patients in control group only receive guideline-directed management in cardiovascular primary or secondary prevention without PCSK9 inhibitor treatment.
  Interventions: Other: Treatment without PCSK9 inhibitors

INTERVENTIONS:
Drug: Treatment with PCSK9 inhibitors — Patients in experimental group are treated with PCSK9 inhibitors (Tafolecimab subcutaneously every two weeks) plus guideline-directed management in cardiovascular primary or secondary prevention.
  Other Names: Treatment with Proprotein convertase subtilisin/kexin type 9 inhibitors
  Arms: Treatment with PCSK9 inhibitors
Other: Treatment without PCSK9 inhibitors — Patients in control group only receive guideline-directed management in cardiovascular primary or secondary prevention without PCSK9 inhibitor treatment.
  Other Names: Treatment without Proprotein convertase subtilisin/kexin type 9 inhibitors
  Arms: Treatment without PCSK9 inhibitors

SUMMARY:
Calcific aortic stenosis (CAS) can cause severe adverse cardiac events, but there are currently no effective drugs that can prevent or delay the progression of the disease. Our trial aims to investigate the effect of PCSK9 inhibitors on preventing or delaying the progression of CAS.

DETAILED DESCRIPTION:
Calcific aortic stenosis (CAS) can cause severe adverse cardiac events, but there are currently no effective drugs that can prevent or delay the progression of the disease. In fact, aortic valve replacement remains the only treatment option. CAS has been shown to be associated with Lp(a), LDL-C and PCSK9. Several observational studies indicated that the use of statins to decrease LDL-C levels was associated with the reduced incidence of CAS, but no randomized controlled trials (RCTs) showd that statins had any benefit on the progression of CAS. This may be related to the limited reduction of LDL-C by statin therapy. The PCSK9 inhibitors have emerged as a new lipid-lowering drug. On the basis of statin therapy, PCSK9 inhibitors can further reduce LDL-C and Lp(a) levels by 50% to 60% and 20% to 30%, respectively. Some studies reported that elevated plasma PCSK9 levels were related to CAS and PCSK9 R46L loss-of-function mutation was associated with lower rates of CAS, and importantly, some observational studies found that PCSK9 inhibitors could reduce the incidence of CAS. Our trial aims to investigate the effect of PCSK9 inhibitors on preventing or delaying the progression of CAS. A total of 160 patients with mild or moderate CAS not currently requiring valve replacement therapy will be enrolled and randomized (stratified by center) in a 1:1 ratio to two groups, the PCSK9 inhibitor treatment group (test group) or the no PCSK9 inhibitor group (control group). All patients will be followed for at least 2 years after randomization. After enrollment, telephone follow-ups will be conducted in the first month and every three months to collect data including medication use, quality-of-life scores, and clinical endpoint events. Doppler echocardiography will be collected at baseline, the 1-year visit, the 2-year visit, and before study withdrawal. Blood samples and aortic computed tomography angiography (CTA) will be collected at baseline, the 2-year visit, and before study withdrawal. The primary endpoint is the annualized mean change in peak aortic jet velocity over the 24-month follow-up period. Secondary endpoints include the annualized mean change in aortic valve area by echocardiography, the annualized mean change in aortic valve calcium score by aortic CTA, the incidence of cardiac valve surgery, and changes in quality-of-life scores. The safety endpoint is a composite of all-cause mortality, non-fatal myocardial infarction, and non-fatal stroke. The results of this trial will provide new insights into the treatment of CAS patients.

Blood samples should be tested for serological indicators, including blood routine, C-reactive protein (CRP), biochemical, coagulation function, brain natriuretic peptide (BNP), markers of myocardial injury, glycosylated hemoglobin, erythrocyte sedimentation rate, cytokines (12 items).

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-85 years old, clinically diagnosed with simple mild or moderate CAVS (echocardiography shows ejection fraction > 50%; valve orifice area > 1.0 cm²; left ventricular stroke volume index > 35 ml/m²; flow velocity ≥ 2 m/s and < 4 m/s, or mean transvalvular pressure gradient < 40 mmHg) and currently not requiring valve replacement therapy;
2. LDL-C ≥ 2.6 and < 4.9 mmol/L, or Lp(a) ≥ 30 mg/dL;
3. Patients who can understand the purpose of the trial, voluntarily participate, sign the informed consent form, and are willing to undergo clinical follow-up in accordance with the trial requirements.

   * The position and method of measurement have been further clarified in ultrasonic measurement to ensure comparability among all enrolled patients, as follows: Aortic valve peak flow velocity, aortic valve mean pressure gradient, and valve orifice area (select images of at least 3 consecutive cardiac cycles with stable heart rate; for atrial fibrillation, select images of more than 5 consecutive cardiac cycles; obtain the peak blood flow velocity of the aortic valve orifice using continuous wave Doppler in the apical 5-chamber view; calculate the instantaneous aortic valve pressure gradient using the simplified Bernoulli equation, and calculate the standardized aortic valve orifice area using the continuity equation; all participating sonographers will receive unified training, perform measurements in fixed views and retain images, which will then be reviewed by two experienced sonographers who are blinded to the trial in the core laboratory).

Exclusion Criteria:

1. Any previous treatment with PCSK9 inhibitors;
2. Patients must be treated with PCSK9 inhibitors by physician's judgment;
3. Patients who cannot maintain PCSK9 inhibitor use for 24 months;
4. Contraindications or hypersensitivity to PCSK9 inhibitors;
5. Suspected or confirmed familial hypercholesterolemia;
6. Fasting triglycerides (TG) >400 mg/dL (4.5 mmol/L) at baseline screening;
7. Thyroid hypofunction;
8. Active or chronic liver disease;
9. Severe renal insufficiency (eGFR <30 mL/min/1.73 m²);
10. History of intracranial hemorrhage;
11. History of alcohol or drug abuse；
12. Known active infection, or severe hematologic, metabolic, or endocrine dysfunction;
13. Systemic corticosteroid or cyclosporine therapy within the past 3 months;
14. Active malignancy;
15. Any life-threatening condition with life expectancy less than 12 months;
16. Rheumatic aortic stenosis;
17. Severe mitral stenosis (mitral valve area <1 cm²);
18. Severe mitral or aortic regurgitation;
19. Planned cardiac valve surgery;
20. Left ventricular ejection fraction < 30% or severe heart failure (NYHA class III or IV);
21. Implanted permanent pacemaker or cardioverter-defibrillator;
22. Drug-refractory arrhythmias;
23. Pregnancy, lactation, or planned pregnancy.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
The annualized mean change in peak aortic jet velocity | Up to 24 months
  The peak aortic jet velocity is measured by echocardiography.

SECONDARY OUTCOMES:
The annualized mean change in aortic valve area | Up to 24 months
  The aortic valve area is measured by echocardiography.
The annualized mean change in aortic valve calcium score | Up to 24 months
  The aortic valve calcification score is measured by aortic computed tomography angiography.
Cardiac valve surgery | Up to 24 months
  Transcatheter aortic valve implantation or surgical aortic valve replacement
Change in quality-of-life scores | Up to 24 months
  Change in quality-of-life scores is assessed with the use of the EQ-5D-3L scale

OTHER OUTCOMES:
Safety endpoint | Up to 24 months
  The safety endpoint is a composite of all-cause mortality, non-fatal myocardial infarction, and non-fatal stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Zhijian Wang, Study Chair — Beijing Anzhen Hospital; Xiaoteng Ma, Principal Investigator — Beijing Anzhen Hospital
Locations (1):
- Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leopold JA. PCSK9 and Calcific Aortic Valve Stenosis: Moving Beyond Lipids. JACC Basic Transl Sci. 2020 Jul 27;5(7):662-664. doi: 10.1016/j.jacbts.2020.06.004. eCollection 2020 Jul. PMID 32760918
- [Background] O'Donoghue ML, Fazio S, Giugliano RP, Stroes ESG, Kanevsky E, Gouni-Berthold I, Im K, Lira Pineda A, Wasserman SM, Ceska R, Ezhov MV, Jukema JW, Jensen HK, Tokgozoglu SL, Mach F, Huber K, Sever PS, Keech AC, Pedersen TR, Sabatine MS. Lipoprotein(a), PCSK9 Inhibition, and Cardiovascular Risk. Circulation. 2019 Mar 19;139(12):1483-1492. doi: 10.1161/CIRCULATIONAHA.118.037184. PMID 30586750
- [Background] Langsted A, Nordestgaard BG, Benn M, Tybjaerg-Hansen A, Kamstrup PR. PCSK9 R46L Loss-of-Function Mutation Reduces Lipoprotein(a), LDL Cholesterol, and Risk of Aortic Valve Stenosis. J Clin Endocrinol Metab. 2016 Sep;101(9):3281-7. doi: 10.1210/jc.2016-1206. Epub 2016 May 24. PMID 27218270
- [Background] Mateos N, Gomez M, Homar A, Garcia-Elias A, Yanez L, Tajes M, Molina L, Ble M, Cladellas M, Roqueta C, Benito B. Plasmatic PCSK9 Levels Are Associated with Very Fast Progression of Asymptomatic Degenerative Aortic Stenosis. J Cardiovasc Transl Res. 2022 Feb;15(1):5-14. doi: 10.1007/s12265-021-10138-4. Epub 2021 Aug 2. PMID 34341879
- [Background] Poggio P, Songia P, Cavallotti L, Barbieri SS, Zanotti I, Arsenault BJ, Valerio V, Ferri N, Capoulade R, Camera M. PCSK9 Involvement in Aortic Valve Calcification. J Am Coll Cardiol. 2018 Dec 18;72(24):3225-3227. doi: 10.1016/j.jacc.2018.09.063. No abstract available. PMID 30545459
- [Background] Raal FJ, Giugliano RP, Sabatine MS, Koren MJ, Langslet G, Bays H, Blom D, Eriksson M, Dent R, Wasserman SM, Huang F, Xue A, Albizem M, Scott R, Stein EA. Reduction in lipoprotein(a) with PCSK9 monoclonal antibody evolocumab (AMG 145): a pooled analysis of more than 1,300 patients in 4 phase II trials. J Am Coll Cardiol. 2014 Apr 8;63(13):1278-1288. doi: 10.1016/j.jacc.2014.01.006. Epub 2014 Feb 5. PMID 24509273
- [Background] Bergmark BA, O'Donoghue ML, Murphy SA, Kuder JF, Ezhov MV, Ceska R, Gouni-Berthold I, Jensen HK, Tokgozoglu SL, Mach F, Huber K, Gaciong Z, Lewis BS, Schiele F, Jukema JW, Pedersen TR, Giugliano RP, Sabatine MS. An Exploratory Analysis of Proprotein Convertase Subtilisin/Kexin Type 9 Inhibition and Aortic Stenosis in the FOURIER Trial. JAMA Cardiol. 2020 Jun 1;5(6):709-713. doi: 10.1001/jamacardio.2020.0728. PMID 32347887
- [Background] Capoulade R, Yeang C, Chan KL, Pibarot P, Tsimikas S. Association of Mild to Moderate Aortic Valve Stenosis Progression With Higher Lipoprotein(a) and Oxidized Phospholipid Levels: Secondary Analysis of a Randomized Clinical Trial. JAMA Cardiol. 2018 Dec 1;3(12):1212-1217. doi: 10.1001/jamacardio.2018.3798. PMID 30476957
- [Background] Capoulade R, Chan KL, Yeang C, Mathieu P, Bosse Y, Dumesnil JG, Tam JW, Teo KK, Mahmut A, Yang X, Witztum JL, Arsenault BJ, Despres JP, Pibarot P, Tsimikas S. Oxidized Phospholipids, Lipoprotein(a), and Progression of Calcific Aortic Valve Stenosis. J Am Coll Cardiol. 2015 Sep 15;66(11):1236-1246. doi: 10.1016/j.jacc.2015.07.020. PMID 26361154
- [Background] Zheng KH, Tsimikas S, Pawade T, Kroon J, Jenkins WSA, Doris MK, White AC, Timmers NKLM, Hjortnaes J, Rogers MA, Aikawa E, Arsenault BJ, Witztum JL, Newby DE, Koschinsky ML, Fayad ZA, Stroes ESG, Boekholdt SM, Dweck MR. Lipoprotein(a) and Oxidized Phospholipids Promote Valve Calcification in Patients With Aortic Stenosis. J Am Coll Cardiol. 2019 May 7;73(17):2150-2162. doi: 10.1016/j.jacc.2019.01.070. PMID 31047003
- [Background] Thanassoulis G, Campbell CY, Owens DS, Smith JG, Smith AV, Peloso GM, Kerr KF, Pechlivanis S, Budoff MJ, Harris TB, Malhotra R, O'Brien KD, Kamstrup PR, Nordestgaard BG, Tybjaerg-Hansen A, Allison MA, Aspelund T, Criqui MH, Heckbert SR, Hwang SJ, Liu Y, Sjogren M, van der Pals J, Kalsch H, Muhleisen TW, Nothen MM, Cupples LA, Caslake M, Di Angelantonio E, Danesh J, Rotter JI, Sigurdsson S, Wong Q, Erbel R, Kathiresan S, Melander O, Gudnason V, O'Donnell CJ, Post WS; CHARGE Extracoronary Calcium Working Group. Genetic associations with valvular calcification and aortic stenosis. N Engl J Med. 2013 Feb 7;368(6):503-12. doi: 10.1056/NEJMoa1109034. PMID 23388002
- [Background] Perrot N, Valerio V, Moschetta D, Boekholdt SM, Dina C, Chen HY, Abner E, Martinsson A, Manikpurage HD, Rigade S, Capoulade R, Mass E, Clavel MA, Le Tourneau T, Messika-Zeitoun D, Wareham NJ, Engert JC, Polvani G, Pibarot P, Esko T, Smith JG, Mathieu P, Thanassoulis G, Schott JJ, Bosse Y, Camera M, Theriault S, Poggio P, Arsenault BJ. Genetic and In Vitro Inhibition of PCSK9 and Calcific Aortic Valve Stenosis. JACC Basic Transl Sci. 2020 Jul 1;5(7):649-661. doi: 10.1016/j.jacbts.2020.05.004. eCollection 2020 Jul. PMID 32760854
- [Background] Guddeti RR, Patil S, Ahmed A, Sharma A, Aboeata A, Lavie CJ, Alla VM. Lipoprotein(a) and calcific aortic valve stenosis: A systematic review. Prog Cardiovasc Dis. 2020 Jul-Aug;63(4):496-502. doi: 10.1016/j.pcad.2020.06.002. Epub 2020 Jun 8. PMID 32526213
- [Background] Youssef A, Clark JR, Koschinsky ML, Boffa MB. Lipoprotein(a): Expanding our knowledge of aortic valve narrowing. Trends Cardiovasc Med. 2021 Jul;31(5):305-311. doi: 10.1016/j.tcm.2020.06.001. Epub 2020 Jun 7. PMID 32525013
- [Background] Capoulade R, Cariou B. Editorial commentary: Lp(a) and calcific aortic valve stenosis: Direct LPA targeting or PCSK9-Lowering therapy? Trends Cardiovasc Med. 2021 Jul;31(5):312-314. doi: 10.1016/j.tcm.2020.06.009. Epub 2020 Jul 2. No abstract available. PMID 32623063
- [Background] Schwartz GG, Steg PG, Szarek M, Bhatt DL, Bittner VA, Diaz R, Edelberg JM, Goodman SG, Hanotin C, Harrington RA, Jukema JW, Lecorps G, Mahaffey KW, Moryusef A, Pordy R, Quintero K, Roe MT, Sasiela WJ, Tamby JF, Tricoci P, White HD, Zeiher AM; ODYSSEY OUTCOMES Committees and Investigators. Alirocumab and Cardiovascular Outcomes after Acute Coronary Syndrome. N Engl J Med. 2018 Nov 29;379(22):2097-2107. doi: 10.1056/NEJMoa1801174. Epub 2018 Nov 7. PMID 30403574
- [Background] Sabatine MS, Giugliano RP, Keech AC, Honarpour N, Wiviott SD, Murphy SA, Kuder JF, Wang H, Liu T, Wasserman SM, Sever PS, Pedersen TR; FOURIER Steering Committee and Investigators. Evolocumab and Clinical Outcomes in Patients with Cardiovascular Disease. N Engl J Med. 2017 May 4;376(18):1713-1722. doi: 10.1056/NEJMoa1615664. Epub 2017 Mar 17. PMID 28304224
- [Background] Seidah NG, Prat A. The Multifaceted Biology of PCSK9. Endocr Rev. 2022 May 12;43(3):558-582. doi: 10.1210/endrev/bnab035. PMID 35552680
- [Background] Punch E, Klein J, Diaba-Nuhoho P, Morawietz H, Garelnabi M. Effects of PCSK9 Targeting: Alleviating Oxidation, Inflammation, and Atherosclerosis. J Am Heart Assoc. 2022 Feb;11(3):e023328. doi: 10.1161/JAHA.121.023328. Epub 2022 Jan 20. PMID 35048716
- [Background] Writing Committee Members; Otto CM, Nishimura RA, Bonow RO, Carabello BA, Erwin JP 3rd, Gentile F, Jneid H, Krieger EV, Mack M, McLeod C, O'Gara PT, Rigolin VH, Sundt TM 3rd, Thompson A, Toly C. 2020 ACC/AHA Guideline for the Management of Patients With Valvular Heart Disease: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. J Am Coll Cardiol. 2021 Feb 2;77(4):e25-e197. doi: 10.1016/j.jacc.2020.11.018. Epub 2020 Dec 17. No abstract available. PMID 33342586
- [Background] Dichtl W, Alber HF, Feuchtner GM, Hintringer F, Reinthaler M, Bartel T, Sussenbacher A, Grander W, Ulmer H, Pachinger O, Muller S. Prognosis and risk factors in patients with asymptomatic aortic stenosis and their modulation by atorvastatin (20 mg). Am J Cardiol. 2008 Sep 15;102(6):743-8. doi: 10.1016/j.amjcard.2008.04.060. Epub 2008 Jul 2. PMID 18774000
- [Background] van der Linde D, Yap SC, van Dijk AP, Budts W, Pieper PG, van der Burgh PH, Mulder BJ, Witsenburg M, Cuypers JA, Lindemans J, Takkenberg JJ, Roos-Hesselink JW. Effects of rosuvastatin on progression of stenosis in adult patients with congenital aortic stenosis (PROCAS Trial). Am J Cardiol. 2011 Jul 15;108(2):265-71. doi: 10.1016/j.amjcard.2011.03.032. Epub 2011 May 10. PMID 21565321
- [Background] Evangelista A, Galian-Gay L, Guala A, Teixido-Tura G, Calvo-Iglesias F, Sevilla T, Bermejo J, Mendez I, Sanchez V, Robledo Carmona JM, Alegret JM, Ferrer-Sistach E, Saura D, Ruiz-Munoz A, Dux-Santoy L, Carmona MA, Huguet M, Cuellar-Calabria H, Sao-Aviles A, Ferreira-Gonzalez I, Rodriguez-Palomares JF. Atorvastatin Effect on Aortic Dilatation and Valvular Calcification Progression in Bicuspid Aortic Valve (BICATOR): A Randomized Clinical Trial. Circulation. 2024 Jun 18;149(25):1938-1948. doi: 10.1161/CIRCULATIONAHA.123.067537. Epub 2024 May 28. PMID 38804148
- [Background] Chan KL, Teo K, Dumesnil JG, Ni A, Tam J; ASTRONOMER Investigators. Effect of Lipid lowering with rosuvastatin on progression of aortic stenosis: results of the aortic stenosis progression observation: measuring effects of rosuvastatin (ASTRONOMER) trial. Circulation. 2010 Jan 19;121(2):306-14. doi: 10.1161/CIRCULATIONAHA.109.900027. Epub 2010 Jan 4. PMID 20048204
- [Background] Rossebo AB, Pedersen TR, Boman K, Brudi P, Chambers JB, Egstrup K, Gerdts E, Gohlke-Barwolf C, Holme I, Kesaniemi YA, Malbecq W, Nienaber CA, Ray S, Skjaerpe T, Wachtell K, Willenheimer R; SEAS Investigators. Intensive lipid lowering with simvastatin and ezetimibe in aortic stenosis. N Engl J Med. 2008 Sep 25;359(13):1343-56. doi: 10.1056/NEJMoa0804602. Epub 2008 Sep 2. PMID 18765433
- [Background] Cowell SJ, Newby DE, Prescott RJ, Bloomfield P, Reid J, Northridge DB, Boon NA; Scottish Aortic Stenosis and Lipid Lowering Trial, Impact on Regression (SALTIRE) Investigators. A randomized trial of intensive lipid-lowering therapy in calcific aortic stenosis. N Engl J Med. 2005 Jun 9;352(23):2389-97. doi: 10.1056/NEJMoa043876. PMID 15944423
- [Background] Nazarzadeh M, Pinho-Gomes AC, Bidel Z, Dehghan A, Canoy D, Hassaine A, Ayala Solares JR, Salimi-Khorshidi G, Smith GD, Otto CM, Rahimi K. Plasma lipids and risk of aortic valve stenosis: a Mendelian randomization study. Eur Heart J. 2020 Oct 21;41(40):3913-3920. doi: 10.1093/eurheartj/ehaa070. PMID 32076698
- [Background] Lincoff AM, Ray KK, Sasiela WJ, Haddad T, Nicholls SJ, Li N, Cho L, Mason D, Libby P, Goodman SG, Nissen SE. Comparative Cardiovascular Benefits of Bempedoic Acid and Statin Drugs. J Am Coll Cardiol. 2024 Jul 9;84(2):152-162. doi: 10.1016/j.jacc.2024.04.048. PMID 38960508
- [Background] Natorska J, Kopytek M, Undas A. Aortic valvular stenosis: Novel therapeutic strategies. Eur J Clin Invest. 2021 Jul;51(7):e13527. doi: 10.1111/eci.13527. Epub 2021 Mar 13. PMID 33621361
- [Background] Rajamannan NM, Evans FJ, Aikawa E, Grande-Allen KJ, Demer LL, Heistad DD, Simmons CA, Masters KS, Mathieu P, O'Brien KD, Schoen FJ, Towler DA, Yoganathan AP, Otto CM. Calcific aortic valve disease: not simply a degenerative process: A review and agenda for research from the National Heart and Lung and Blood Institute Aortic Stenosis Working Group. Executive summary: Calcific aortic valve disease-2011 update. Circulation. 2011 Oct 18;124(16):1783-91. doi: 10.1161/CIRCULATIONAHA.110.006767. No abstract available. PMID 22007101
- [Background] Genereux P, Stone GW, O'Gara PT, Marquis-Gravel G, Redfors B, Giustino G, Pibarot P, Bax JJ, Bonow RO, Leon MB. Natural History, Diagnostic Approaches, and Therapeutic Strategies for Patients With Asymptomatic Severe Aortic Stenosis. J Am Coll Cardiol. 2016 May 17;67(19):2263-2288. doi: 10.1016/j.jacc.2016.02.057. Epub 2016 Apr 2. PMID 27049682
- [Background] Lindman BR, Dweck MR, Lancellotti P, Genereux P, Pierard LA, O'Gara PT, Bonow RO. Management of Asymptomatic Severe Aortic Stenosis: Evolving Concepts in Timing of Valve Replacement. JACC Cardiovasc Imaging. 2020 Feb;13(2 Pt 1):481-493. doi: 10.1016/j.jcmg.2019.01.036. Epub 2019 Jun 12. PMID 31202751
- [Background] Yang Y, Wang Z, Chen Z, Wang X, Zhang L, Li S, Zheng C, Kang Y, Jiang L, Zhu Z, Gao R. Current status and etiology of valvular heart disease in China: a population-based survey. BMC Cardiovasc Disord. 2021 Jul 13;21(1):339. doi: 10.1186/s12872-021-02154-8. PMID 34256700
- [Background] Lindman BR, Clavel MA, Mathieu P, Iung B, Lancellotti P, Otto CM, Pibarot P. Calcific aortic stenosis. Nat Rev Dis Primers. 2016 Mar 3;2:16006. doi: 10.1038/nrdp.2016.6. PMID 27188578
- [Background] Otto CM, Newby DE, Hillis GS. Calcific Aortic Stenosis: A Review. JAMA. 2024 Dec 17;332(23):2014-2026. doi: 10.1001/jama.2024.16477. PMID 39527048